CLINICAL TRIAL: NCT00798642
Title: National Center for Complementary & Alternative Medicine, The Role of Gut-Directed Hypnotherapy in Relapse Prevention for Ulcerative Colitis
Brief Title: Ulcerative Colitis Relapse Prevention Trial, Hypnosis
Acronym: UCRPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Laurie Keefer, Associate Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R21AT003204 (NIH); R21AT003204 (NIH)
Record Dates: First submitted 2008-11-25; First posted 2008-11-26 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2014-04

CONDITIONS: Ulcerative Colitis; Inflammatory Bowel Disease
Keywords: Hypnotherapy; Ulcerative Colitis; Inflammatory Bowel Disease; Gastrointestinal Diseases; Digestive System Diseases; Intestinal Diseases; Colonic Diseases
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases; Gastrointestinal Diseases; Digestive System Diseases; Intestinal Diseases; Colonic Diseases | interventions — Hypnosis; Standard of Care; Mind-Body Therapies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Hypnotherapy (Active Comparator)
  Interventions: Behavioral: Hypnotherapy
- Standard care (Placebo Comparator)
  Interventions: Behavioral: Standard care
- Mind Body Therapy (Placebo Comparator)
  Interventions: Behavioral: Mind Body Therapy

INTERVENTIONS:
Behavioral: Hypnotherapy — 8 weeks of gut-directed hypnotherapy
  Other Names: HYP
  Arms: Hypnotherapy
Behavioral: Standard care — 8 weeks of standard of care
  Other Names: SC
  Arms: Standard care
Behavioral: Mind Body Therapy — 8 weeks of mind-body therapy
  Other Names: MB
  Arms: Mind Body Therapy

SUMMARY:
The UCRPT is a randomized controlled trial to determine if a type of hypnotherapy will maintain remission in patients affected by Ulcerative Colitis.

DETAILED DESCRIPTION:
The purpose of the study is to determine whether hypnotherapy can serve as an effective therapy for patients with Ulcerative Colitis (UC), a chronic, relapsing and remitting inflammatory bowel disease (IBD).

The goal of this study is to determine if mind-body therapy is an effective complementary therapy for IBD, meaning a therapy to be used in conjunction with your standard treatment provided by your gastroenterologist. Standard treatment for UC often includes a combination approach and may include medications such as mesalamine, corticosteroids or immunomodulators. Mind-body therapy or hypnosis has been used to reduce stress and subsequent disease activity in patients with gastrointestinal diseases including IBD and Irritable Bowel Syndrome. It has also been shown to improve immune function and reduce inflammation in other health conditions such as cancer and arthritis.

In this study, patients with inactive UC will be randomized to one of three groups. Two groups will undergo one of two mind-body therapies, which may include relaxation techniques or other techniques aimed at identifying the impact of UC on your psyche along with standard care for their UC. The other group will undergo 8 weeks of standard care without mind-body therapy. Clinical assessment measures will be repeated at 8 weeks, 12 weeks, 24 weeks and 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* male and female patients between the ages of 18 and 70 of any ethnicity
* endoscopy-confirmed (within the past 2 years) mild or moderately severe Ulcerative Colitis (at time of previous flare)
* inactive disease at the time of recruitment:
* Mayo score <2 with no subscale >1
* no rectal bleeding
* Physician Global Assessment Score (PGA) = 0
* 2 weeks of baseline daily symptom diaries that support criteria for inactive disease
* documented disease flare within the past 1.5 years to enhance the opportunity to observe differences between groups in a 1-year trial .
* no medication or a stable dose of maintenance medication (i.e. mesalamine or sulfasalazine) for at least one month prior to enrollment.
* If taking maintenance medication: an increase in dose will be considered a relapse
* If taking no medication: initiation of any medication will be considered a relapse

Exclusion Criteria:

* active disease
* daily rectal bleeding for past 7 days
* Mayo Score > 2, any subscale > 1
* PGA score >0
* history of severe or fulminant UC
* most recent flare included > 6 bloody stools a day
* history of of toxicity including fever, tachycardia, anemia or an elevated Erythrocyte sedimentation rate (ESR) ∙ history of continuous bleeding, blood transfusion requirement, abdominal tenderness and distension, and colonic dilation on abdominal plain films
* other gastrointestinal conditions
* Crohn's Disease (CD)
* short-bowel syndrome
* celiac sprue
* irritable bowel syndrome (IBS)
* renal or hepatic disease
* positive stool exam (bacteria, ova, parasites)
* C-difficile
* history of colon resection
* steroid-dependent, patients taking oral steroids within the past 30 days, topical steroids within the past week, quit smoking in the past 30 days given the known effects of smoking cessation on UC disease flare 23.
* contraindications for hypnotherapy
* unresolved history of physical or sexual abuse
* a current or past dissociative disorder (i.e. Borderline PD, PTSD)
* history of psychosis (including mania)
* history of psychiatric hospitalization, including for self-harm or SI/HI
* current substance abuse
* severe psychiatric disorder
* patients who are resistant to hypnosis as a result of religious or moral beliefs or any other reason

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2007-07; Primary Completion 2011-11 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
feasibility | 52 weeks

SECONDARY OUTCOMES:
Estimated effect sizes | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Laurie Keefer, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Feinberg School of Medicine, Chicago, Illinois, United States

REFERENCES:
- [Derived] Tiles-Sar N, Neuser J, de Sordi D, Baltes A, Preiss JC, Moser G, Timmer A. Psychological interventions for treatment of inflammatory bowel disease. Cochrane Database Syst Rev. 2025 Apr 17;4(4):CD006913. doi: 10.1002/14651858.CD006913.pub3. PMID 40243391
- [Derived] Keefer L, Taft TH, Kiebles JL, Martinovich Z, Barrett TA, Palsson OS. Gut-directed hypnotherapy significantly augments clinical remission in quiescent ulcerative colitis. Aliment Pharmacol Ther. 2013 Oct;38(7):761-71. doi: 10.1111/apt.12449. Epub 2013 Aug 19. PMID 23957526